CLINICAL TRIAL: NCT03514875
Title: Effects of Mitochondrial-targeted Antioxidant on Carotid Artery Endothelial Function and Brain Blood Flow in Mild Cognitive Impairment (MCI) Patients
Brief Title: Effects of Mitochondrial-targeted Antioxidant on Mild Cognitive Impairment (MCI) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: discontinued due to change in operating plans prior to study initiation and enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0088-18-FB
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease, Early Onset; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized, cross-over design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ-Placebo (Experimental): Subjects will be tested on two different days, first day will be baseline and MitoQ intake, and second day will be placebo intake. Testing will take place 40-minutes after MitoQ and placebo intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: MitoQ; Dietary Supplement: Placebo
- Placebo-MitoQ (Experimental): Subjects will be tested on two different days, first day will be baseline and placebo intake, and second day will be MitoQ intake. Testing will take place 40-minutes after placebo and MitoQ intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: MitoQ; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ is a mitochondria-targeting antioxidant, which should improve NO bioavailability, and therefore vasodilation
Dietary Supplement: Placebo — A placebo will be used in a double blinded, randomized, cross-over design

SUMMARY:
Neurodegenerative diseases such as Mild Cognitive Impairment, Alzheimer's, and dementia affect millions of Americans. Although these diseases are heavily researched, there is very little research examining the impact of attenuated carotid artery endothelial function and cerebrovascular blood flow on cognitive function. This is surprising, as cerebrovascular oxygenation has been shown to be strongly associated with reduced cognitive function and the pathogenesis of neurodegenerative diseases. For example, hypertension, diabetes, and high cholesterol have been shown to increase the risk of Alzheimers related dementia. Therefore, the purpose of this proposed study will be to examine the effects of MitoQ supplementation on carotid artery vasodilatory function and cerebrovascular blood flow in those suffering from Mild Cognitive Impairment (MCI). MitoQ is a mitochondria-targeting antioxidant that can improve nitric oxide production in the blood vessel, which should improve endothelial function, and thus cerebrovascular blood flow.

DETAILED DESCRIPTION:
Metabolic disease parameters, such as hyperlipidemia and hypertension have been observed in Alzheimer's disease and dementia. The causes of neurodegenerative diseases like Alzheimers are not completely understood. However, increasing amounts of evidence are pointing to vascular dysfunction as a cause of this disease. Known as the vascular hypothesis, pathology is suggested to begin with cerebral hypoperfusion through attenuated blood flow via clogged carotid arteries. Hypoperfusion of cerebral cells means that they do not receive enough oxygen to function optimally. This lack of oxygen is believed to lead to cognitive impairment. It is hypothesized that these metabolic conditions can damage the endothelial wall, leading to impaired vasodilation and blood flow. This damage occurs in the carotid arteries, which would limit blood flow to the brain. This impaired blood flow also results from higher levels of reactive oxygen species (ROS), which reduce the bioavailability of nitric oxide (NO), an important vasodilator. Antioxidants, such as MitoQ, reduce these ROS and thus increase the NO availability, which improves endothelial function. This study will measure the use of the antioxidant MitoQ to reduce this endothelial dysfunction, thereby improving blood flow in the carotid arteries. Blood vessel health can be measured by how much bigger or smaller a vessel can become, because the ability of the vessel to change size is very important to make sure that blood is delivered to the tissues of the body. This study is being done to help us understand if endothelial dysfunction in Mild Cognitive Impairment (MCI) patients leads to the pathogenesis of the disease.

We will examine how endothelial function and cerebrovascular blood flow changes after consumption of MitoQ. We hope to achieve this through measures of carotid artery blood flow and brachial artery blood flow, using a doppler ultrasound for both, while using flow mediated dilation when measuring the brachial artery. The flow-mediated dilation test is a validated and safe assessment of endothelial function and vascular health. The premise behind the assessment is that endothelium produces autocoids, like nitric oxide, that dilate in response to shear stress. Flow-mediated dilation has been shown to be an effective tool to assess endothelial function in the peripheral and coronary vasculature. This assessment of endothelial health can be used in healthy individuals to detect risk for cardiovascular disease. We will also utilize near infrared spectroscopy to measure tissue oxygenation in the brain, which is also a measure of improved blood flow, and will measure brain neural activity with an EEG. Finally, we will collect blood samples to measure the change in ROS levels before and after MitoQ consumption

ELIGIBILITY:
Inclusion Criteria:

1. be able to give written, informed consent
2. Have a clinical diagnosis of Mild Cognitive Impairment (MCI) verified by a medical doctor
3. have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks.
4. Free of kidney, metabolic or cardiovascular disease, including hypertension (stage 2) and previous cardiac events
5. be between 50-85 years old

Exclusion Criteria:

1. All participants must be free from smoking and alcohol abuse
2. Not be taking prescription drugs (other than oral contraceptives, blood pressure lowering drugs, and metformin)
3. Must not be diagnosed with Alzheimer's disease.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Carotid artery blood flow | 2 Days
  Blood flow in the carotid artery will be measured with ultrasound

SECONDARY OUTCOMES:
Oxidative Stress | 2 days
  Blood draws will be taken to measure oxidative stress markers in the blood
Cerebrovascular Oxygenation | 2 Days
  Near-infrared spectroscopy will be used to measure cerebrovascular oxygenation
Brain Electrical Activity | 2 Days
  EEG will measure brain electrical activity
Endothelial Function | 2 Days
  Flow-mediated dilation will be used to measure vasodilation in the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Song-young Park, PhD, Principal Investigator — University of Nebraska

REFERENCES:
- [Background] Kelleher RJ, Soiza RL. Evidence of endothelial dysfunction in the development of Alzheimer's disease: Is Alzheimer's a vascular disorder? Am J Cardiovasc Dis. 2013 Nov 1;3(4):197-226. PMID 24224133
- [Background] Luchsinger JA, Reitz C, Honig LS, Tang MX, Shea S, Mayeux R. Aggregation of vascular risk factors and risk of incident Alzheimer disease. Neurology. 2005 Aug 23;65(4):545-51. doi: 10.1212/01.wnl.0000172914.08967.dc. PMID 16116114
- [Background] Green DJ, Jones H, Thijssen D, Cable NT, Atkinson G. Flow-mediated dilation and cardiovascular event prediction: does nitric oxide matter? Hypertension. 2011 Mar;57(3):363-9. doi: 10.1161/HYPERTENSIONAHA.110.167015. Epub 2011 Jan 24. PMID 21263128
- [Background] Green DJ, Dawson EA, Groenewoud HM, Jones H, Thijssen DH. Is flow-mediated dilation nitric oxide mediated?: A meta-analysis. Hypertension. 2014 Feb;63(2):376-82. doi: 10.1161/HYPERTENSIONAHA.113.02044. Epub 2013 Nov 25. PMID 24277765